CLINICAL TRIAL: NCT05330468
Title: Regent China Post-Market Clinical Follow-up Study
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10412
Record Dates: First submitted 2022-04-13; First posted 2022-04-15 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-09

CONDITIONS: Valvular Heart Disease; Aortic Valve Disease
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Abbott Regent MHV: Subjects implanted with an Abbott Regent MHV replacement of the aortic valve.
  Interventions: Device: Abbott Mechanical Heart Valve (MHV) Regent™

INTERVENTIONS:
Device: Abbott Mechanical Heart Valve (MHV) Regent™ — SJM Regent™- Standard cuff (Model number AGN-751); SJM Regent™- FlexCuff™ (Model number AGFN-756)

SUMMARY:
Regent China Post-Market Clinical Follow-Up (RC-PMCF): this clinical study is to confirm the safety and performance of Abbott's Regent MHV for replacement of native or prosthetic aortic valves in a Chinese population.

DETAILED DESCRIPTION:
The purpose of the RC-PMCF study is to meet the post-market clinical followup (PMCF) requirements of the National Medical Products Administration (NMPA). The primary objective of this clinical study is to confirm the safety and performance of Abbott's Regent MHV for replacement of native or prosthetic aortic valves in a Chinese population. This is a prospective, observational, multi-center study of subjects clinically indicated for implantation of an Abbott Medical's Regent Valve.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is eligible to be implanted with Regent to replace a native or prosthetic aortic valve per Regent's IFU.
2. Subject will be >18 years of age at time of being consented.
3. Subject, provides written informed consent prior to any clinical investigation-specific procedure.

Exclusion Criteria:

1. Subject is unable to tolerate anticoagulation therapy.
2. Subject has active endocarditis.
3. Subject is currently participating in another clinical investigation which may interfere with the effectiveness of anticoagulation therapy.
4. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period. Women of child-bearing potential must have a documented negative pregnancy test within one week prior to enrollment.
5. Subject has anomalous anatomy or medical, surgical, psychological or social history or conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements of the clinical investigation results.
6. Subject is unable to read or write or has a mental illness or disability that impairs their ability to provide written informed consent.
7. Subject's life expectancy is less than 1 year in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This clinical investigation will enroll male and female subjects who will be undergoing replacement of a native or prosthetic aortic heart valve. Patients must meet all general eligibility criteria and provide written informed consent prior to sites conducting any investigation-specific procedures not considered standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Brunner, Study Director — Abbott
Locations (5):
- China (5):
  - The People's Hospital of Gaozhou, Gaozhou
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - Wuhan Union Hospital of China, Wuhan
  - Affiliated Hospital of Zunyi Medical University, Zunyi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 200 subjects were enrolled across 5 investigational sites between 2022 and 2023. Each subject received a Regent MHV implant. Abbott obtained agreement from the Regulatory Bodies to reduce the follow-up period to one year. The final subject follow-up visit occurred in October of 2024.
Period: Overall Study
Arm/Group | Abbott Regent MHV
Started | 200
Completed | 186
Not Completed | 14
Not completed — Death | 6
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Abbott Regent MHV
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 107
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 200
Aortic Regurgitation [Count of Participants; unit: Participants] | 167

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint: The Freedom From Valve-related Mortality
Description: Valve-related mortality is any death caused by structural valve deterioration, nonstructural dysfunction, valve thrombosis, embolism, bleeding event, or operated valve endocarditis; death related to reintervention on the operated valve; or sudden, unexplained death. Deaths caused by heart failure in patients with advanced myocardial disease and satisfactorily functioning cardiac valves are not counted. Specific causes of valve-related deaths should be reported.
Time Frame: At one year
Population: The analysis population included all subjects who provided written informed consent and underwent an implant of a Regent MHV device.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abbott Regent MHV
Number analyzed (Participants) | 200
percentage of participants | 98.4 [95.2 to 99.5]

2. Primary Outcome: Primary Performance Endpoint: The Freedom From Valve-related Reoperation
Description: Valve-related reoperation includes any reintervention that is a surgical or percutaneous interventional catheter procedure that repairs, otherwise alters or adjusts, or replaces the previously implanted prosthesis or repaired valve.
Time Frame: At one year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abbott Regent MHV
Number analyzed (Participants) | 200
percentage of participants | 99.5 [96.3 to 99.9]

ADVERSE EVENTS:
Time Frame: At one year
Arm/Group | Abbott Regent MHV
All-Cause Mortality (participants affected / at risk) | 6/200
Serious Adverse Events (participants affected / at risk) | 67/200
Other Adverse Events (participants affected / at risk) | 10/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abbott Regent MHV (N=200)
Coagulopathy (Blood and lymphatic system disorders) | 2
Arrhythmia (Cardiac disorders) | 4
Atrial Fibrillation (Cardiac disorders) | 1
Atrioventricular Block Complete (Cardiac disorders) | 1
Cardiac Failure (Cardiac disorders) | 4
Cardiac Tamponade (Cardiac disorders) | 1
Cardiogenic Shock (Cardiac disorders) | 1
Cardiorenal Syndrome (Cardiac disorders) | 1
Low Cardiac Output Syndrome (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 2
Ventricular Fibrillation (Cardiac disorders) | 2
Inguinal Hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest Discomfort (General disorders) | 1
Death (General disorders) | 1
Impaired Healing (General disorders) | 1
Paravalvular Regurgitation (General disorders) | 1
Pyrexia (General disorders) | 1
Fungal Infection (Infections and infestations) | 1
Infection (Infections and infestations) | 4
Periodontitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia Bacterial (Infections and infestations) | 1
Postoperative Wound Infection (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Foreign Body in Gastrointestinal Tract (Injury, poisoning and procedural complications) | 1
Coagulation Test Abnormal (Investigations) | 2
International Normalised Ratio Increased (Investigations) | 1
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Ischemic Stroke (Nervous system disorders) | 1
Calculus Urinary (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal Cyst (Renal and urinary disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 1
Arterial Insufficiency (Vascular disorders) | 1
Hemorrhage (Vascular disorders) | 7
Vasculitis Necrotising (Vascular disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abbott Regent MHV (N=200)
Aortic Valve Incompetence (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 2
Atrial Fibrillation (Cardiac disorders) | 1
Atrial Flutter (Cardiac disorders) | 1
Cardiac Failure (Cardiac disorders) | 1
Chest Discomfort (General disorders) | 1
Ischaemic Stroke (Nervous system disorders) | 2
Transient Ischaemic Attack (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restrictions on the PI is that 1) following the earliest of (i) the sponsor's trial results disclosure; or (ii) twelve months after study completion/termination at all study sites, the PI shall publish trial results; 2) the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is equal to or more than 60 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT05330468/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT05330468/SAP_001.pdf